CLINICAL TRIAL: NCT04314999
Title: Häufigkeit Der Infestation Mit Parasiten Bei Patienten Mit Chronisch Spontaner Urtikaria, Eine Retrospektive Datenanalyse
Brief Title: Frequency of Parasite Infestation in Patients With Chronic Spontaneous Urticaria
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01953;sp20Steveling2
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Chronic Spontaneous Urticaria; Parasitic Disease
Keywords: Chronic Spontaneous Urticaria; Parasitic disease
MeSH Terms: conditions — Chronic Urticaria; Parasitic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with a chronic spontaneous urticaria: Patients with a chronic spontaneous urticaria who were being treated at the allergology of the university hospital Basel between the 1st of June and the 30th of September
  Interventions: Diagnostic Test: Examination of stool samples

INTERVENTIONS:
Diagnostic Test: Examination of stool samples — Tests for diagnosis of parasitic diseases

SUMMARY:
The goal of this study is to describe the prevalence and the type of parasite in patients with a chronic spontaneous urticaria as well as to describe the associations between parasitic disease and the characteristics of the patients, for example eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a chronic spontaneous urticaria
* Age: 17 years old and up

Exclusion Criteria:

* No diagnosis of a chronic spontaneous urticaria
* Age: younger than 17 years

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a chric spontaneous urticaria who were being treated at the allergology of the university hospital Basel between the 1st of June and the 30th of September.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with parasite infestation | Patients with a chronic spontaneous urticaria that were treated at the University hospital basel between the 1st of June 2019 and the 30th of September 2019
  assess number of patients with chronic spontaneous urticaria that have a parasite infestation (Analysis of stool samples by the Swiss Tropical and Public Health Institute (TPH), Basel)
Most common parasite subgroup | Patients with a chronic spontaneous urticaria that were treated at the University hospital basel between the 1st of June 2019 and the 30th of September 2019
  subtype determination from stool samples was performed by the Swiss TPH, Basel by polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Correlation between migration Background/ travel history of the patients and parasite infestation | Patients with a chronic spontaneous urticaria that were treated at the University hospital basel between the 1st of June 2019 and the 30th of September 2019
  examine travel history and migration background of patients
Correlation between gastrointestinal complaints of the patients and parasite infestation | Patients with a chronic spontaneous urticaria that were treated at the University hospital basel between the 1st of June 2019 and the 30th of September 2019
  anamnesis of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Esther Steveling-Klein, Dr. med., Principal Investigator — Allergology, University Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland